

### TRIAL STATISTICAL ANALYSIS PLAN

c26502649-01

**BI Trial No.:** 1371-0004

**Title:** Relative bioavailability of a single oral dose of BI 894416 when

administered alone or in combination with multiple oral doses of itraconazole in healthy male subjects (an open-label, one-way

crossover study)

Including Protocol Amendments 1 and 2 [c24667886-03]

Investigational

**Product(s):** 

BI 894416

Responsible trial statistician(s):

Phone:

Fax:

Final

Date of statistical

analysis plan:

06-FEB-2019 SIGNED

Version:


Proprietary confidential information

 ${\small ©~2019~Boehringer~Ingelheim~International~GmbH~or~one~or~more~of~its~affiliated~companies.~All~rights~reserved.}$ 

This document may not - in full or in part - be passed on, reproduced, published or otherwise used without prior written permission.

**7.8.1** 

TSAP for BI Trial No: 1371-0004 

Proprietary confidential information © 2019 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

| 1. | TA | BLE | $\mathbf{OE}$ | CON | TEN | TC |
|----|----------------|------|---------------|-----|-----|-----|
| 1. | $\mathbf{I} P$ | ADLL | <b>U</b> F | CUN | | 110 |

| TITLE I | PAGE | 1 |
|---|---|---|
| 1. | TABLE OF CONTENTS. | 2 |
| LIST OF | TABLES | |
| | LIST OF ABBREVIATIONS | |
| 2. | | |
| 3. | INTRODUCTION | 7 |
| 4. | CHANGES IN THE PLANNED ANALYSIS OF THE STUDY | 8 |
| 5. | ENDPOINTS | 9 |
| 5.1 | PRIMARY ENDPOINTS | 9 |
| 5.2 | SECONDARY ENDPOINTS | |
| 5.2.1<br>5.2.2 | Key secondary endpoint | |
| 6.<br>6.1<br>6.2 | GENERAL ANALYSIS DEFINITIONSTREATMENTSIMPORTANT PROTOCOL DEVIATIONS | 11 |
| 6.3 | SUBJECT SETS ANALYSED | |
| 6.5 | POOLING OF CENTRES | 13 |
| 6.6 | HANDLING OF MISSING DATA AND OUTLIERS | |
| <b>6.7</b> | BASELINE, TIME WINDOWS AND CALCULATED VISITS | 13 |
| <b>7.</b> | PLANNED ANALYSIS | 15 |
| <b>7.1</b> | DEMOGRAPHIC AND OTHER BASELINE CHARACTERISTICS | |
| 7.2 | CONCOMITANT DISEASES AND MEDICATION | |
| 7.3 | TREATMENT COMPLIANCE | |
| 7.4<br>7.5 | PRIMARY ENDPOINT SECONDARY ENDPOINTS | |
| 7.5.1 | Key secondary endpoint | |
| 7.5.2 | Secondary endpoints | |
| 7.7 | EXTENT OF EXPOSURE | |
| <b>7.8</b> | SAFETY ANALYSIS | 18 |

| TSAP | for BI | <b>Trial No:</b> | 1371- | -0004 |
|------|--------|------------------|-------|-------|
|------|--------|------------------|-------|-------|


| Proprietar | ry confidential information © 2019 Boehringer Ingelheim International Gn | nbH or one or more of its affiliated companies |
|---|---|---|
| 7.8.2 | Laboratory data | 19 |
| 7.8.3 | Vital signs | 20 |
| 7.8.4 | Others | 20 |
| 8. | REFERENCES | 21 |
| 10. | HISTORY TABLE | 27 |

| TSAP | for BI | Trial N | o: 13 | 71-0004 |
|------|--------|---------|-------|---------|
|------|--------|---------|-------|---------|

TSAP for BI Trial No: 1371-0004 

Proprietary confidential information © 2019 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

# LIST OF TABLES

| Table 6.1: 1 Analysis phases for statistical analysis of AEs | |
|--------------------------------------------------------------|----|
| | .1 |
| Table 10: 1 History table | |

TSAP for BI Trial No: 1371-0004 

Proprietary confidential information © 2019 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

#### 2. LIST OF ABBREVIATIONS

| Term | Definition / description |
|---|---|
| AE | Adverse Event |
| AESI | Adverse event of special interest |
| ALT | Alanine aminotransferase |
| ANOVA | Analysis of variance |
| AST | Aspartate aminotransferase |
| $\mathrm{AUC}_{0	ext{-tz}}$ | Area under the concentration-time curve of the analyte in plasma over the time interval from 0 to the last quantifiable data point |
| $\mathrm{AUC}_{0\text{-}\infty}$ | Area under the concentration-time curve of the analyte in plasma from $0$ to infinity |
| BI | Boehringer Ingelheim |
| BP | Blood pressure |
| $C_{\text{max}}$ | Maximum measured concentration of the analyte in plasma |
| CTP | Clinical Trial Protocol |
| CTR | Clinical Trial Report |
| CV | Arithmetic coefficient of variation |
| ECG | Electrocardiogram |
| gCV | geometric coefficient of variation |
| gMean | Geometric mean |
| ICH | International Conference On Harmonisation |
| IPD | Important protocol deviations |
| IQRMP | Integrated quality and risk management plan |
| ITZ | Itraconazole |
| MedDRA | Medical Dictionary For Regulatory Activities |
| PK | Pharmacokinetics |
| PKS | Pharmacokinetic parameter set |
| PR | Pulse rate |
| RAGe | Report appendix generator |
| RPM | Report Planning Meeting |
| SAE | Serious adverse event |
| SD | Standard Deviation |
| SOC | System Organ Class |

TSAP for BI Trial No: 1371-0004 

Proprietary confidential information © 2019 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

| Term | Definition / description |
|------|---------------------------------|
| TS | Treated set |
| TSAP | Trial Statistical Analysis Plan |
| ULN | Upper limit of normal range |

TSAP for BI Trial No: 1371-0004

Proprietary confidential information © 2019 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

#### 3. INTRODUCTION

As per ICH E9 (1), the purpose of this document is to provide a more technical and detailed elaboration of the principal features of the analysis described in the revised CTP, and to include detailed procedures for executing the statistical analysis of the primary and secondary variables and other data.

This TSAP assumes familiarity with the CTP and its amendments. In particular, the TSAP is based on the planned analysis specification as written in CTP Section 7 "Statistical Methods and Determination of Sample Size". Therefore, TSAP readers may consult the revised CTP for more background information on the study, e.g., on study objectives, study design and population, treatments, definition of measurements and variables, planning of sample size, randomisation.

Study data will be stored in a trial database within the Oracle Clinical<sup>TM</sup> system.

The statistical analyses will be performed within the validated working environment CARE, including SAS<sup>TM</sup> (current Version 9.4, by SAS Institute Inc., Cary, NC, USA), and a number of SAS<sup>TM</sup>-based tools (e.g., macros for the analyses of AE data or laboratory data; Report Appendix Generator system (RAGe) for compilation/formatting of the CTR appendices).

PK parameters will be calculated using Phoenix WinNonlin<sup>TM</sup> software (version Phoenix 6.3, Certara USA Inc., Princeton, NJ, USA).

#### CHANGES IN THE PLANNED ANALYSIS OF THE STUDY 4.

All analyses described in this TSAP are in accordance with the statistical methods described in the revised CTP.

### 5. ENDPOINTS

#### 5.1 PRIMARY ENDPOINTS

Primary endpoints are PK endpoints of BI 894416 as defined in Section 2.1.2 of the CTP:

- $AUC_{0-tz}$  (area under the concentration-time curve of the analyte in plasma over the time interval from 0 to the last quantifiable data point)
- $C_{max}$  (maximum measured concentration of the analyte in plasma)

#### 5.2 SECONDARY ENDPOINTS

### 5.2.1 Key secondary endpoint

Not applicable.

## 5.2.2 Secondary endpoint

Secondary endpoint of this trial is  $AUC_{0-\infty}$  of BI 894416 in plasma, as defined in Section 2.1.3 of the CTP.

TSAP for BI Trial No: 1371-0004 

Proprietary confidential information © 2019 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

TSAP for BI Trial No: 1371-0004 Proprietary confidential information © 2019 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

#### 6. **GENERAL ANALYSIS DEFINITIONS**

#### 6.1 **TREATMENTS**

For basic study information on treatments to be administered, assignment of treatment groups, and selection of doses, cf. Section 4 of the CTP.

Each subject is planned to be treated in two subsequent treatment periods. In the first treatment period, subjects will receive a single dose of 3 mg of BI 894416 (reference treatment). In the second treatment period, subjects will receive treatment with itraconazole 200 mg once daily over 5 days together with an administration of a single dose of 3 mg of BI 894416 on the fourth day of itraconazole treatment (test treatment). The sequence of these treatment periods is fixed and the same for all subjects.

For statistical analyses of AEs, the following separate analysis phases will be defined for each subject:

| Table 6.1: 1 | Analysis 1 | phases f | or statistical | analysis o | of AEs |
|--------------|------------|----------|----------------|------------|--------|

| Study analysis phase | Label | Start | End |
|---|---|---|---|
| Screening | Screening | Date of informed consent | Date/time of first administration of BI 894416 |
| On treatment<br>BI 894416 | BI | Date/time of first administration of BI 894416 | Date/time of first administration of itraconazole |
| On treatment ITZ | ITZ | Date/time of first administration of itraconazole | Date/time of second administration of BI 894416 |
| On treatment<br>BI 894416 +<br>ITZ | BI + ITZ | Date/time of second administration of BI 894416 | 12:00 a.m. on day after subject's trial termination date |

CTR Section 15, Appendix 16.1.13.1.8.2 and Appendix 16.1.13.1.8.3 AE displays will present results for the on-treatment phase only.

In CTR Section 15 AE tables (but not in Appendix 16.1.13.1.8.2 and Appendix 16.1.13.1.8.3 AE tables), the following totals will be provided in addition:

- "Total BI", defined as the total over all on-treatment phases involving BI
- "Total on-trt", defined as the total over all on-treatment phases

CTR Appendix 16.1.13.1.8.1 displays will present results for the screening and on-treatment phases.

Additionally to the totals defined above, the following total will be provided in CTR Section 16.1.13.1.8.1 AE tables:

"Total", defined as the total over all study phases (screening + on-treatment)

Statistical analyses of safety laboratory tests and vital signs will be conducted by treatment period (BI vs. BI+ITZ).

More details on the technical implementation of these analyses are provided in the ADS Plan of this TSAP.

#### 6.2 IMPORTANT PROTOCOL DEVIATIONS

Consistency check listings (for identification of deviations from time windows) and a list of protocol deviations (e.g. deviations in drug administration, in blood sampling times, etc.) will be provided to be discussed at the RPM/DBLM. At this meeting, it will be decided whether a discrepant data value can be used in analyses or whether it must be corrected in the clinical database. Each protocol deviation must be assessed to determine whether it is an IPD. For definition of IPDs, and for the process of identification of these, refer to the BI reference document "Identify and Manage Important Protocol Deviations (iPD)" (2).

If any IPDs are identified, they are to be summarised into categories and will be captured in the RPM/DBLM minutes. Categories which are considered to be IPDs in this trial are defined in the integrated quality and risk management plan (IQRMP). If the data show other IPDs, the definition in the IQRMP will be supplemented accordingly by the time of the RPM/DBLM.

IPDs will be summarised and listed.

#### 6.3 SUBJECT SETS ANALYSED

All entered subjects who received study medication will be included in the safety analysis and in the PK analysis depending on the availability of measurement values, and on their adherence to the CTP.

The following subject sets will be defined for statistical analysis:

- Treated set (TS):
  - This subject set includes all subjects who received at least one dose of study drug. This is the full analysis set population in the sense of ICH-E9 (1). It will be used for analysis of safety, demographic data and baseline characteristics.
- Pharmacokinetic parameter set (PKS):
  This subject set includes all subjects in the TS who provide at least one PK parameter that was not excluded because of IPDs relevant to the statistical evaluation of PK endpoints as defined in Section 7.3 of the CTP.

The discussion of all exceptional cases and problems and the decisions on the allocation of subjects to analysis sets will be made at latest at the RPM/DBLM.

Table 6.3: 1 Subject sets analysed

TSAP for BI Trial No: 1371-0004

| | Sub | ject set |
|--------------------------------|-----|----------|
| Class of endpoint | TS | PKS |
| Disposition | X | |
| Exposure | X | |
| IPDs | X | |
| Demographic/baseline endpoints | X | |
| Safety parameters | X | |
| Primary endpoints | | X |
| Secondary endpoint | | X |
| Further PK endpoints | | X |

#### 6.5 POOLING OF CENTRES

This section is not applicable, because the study was performed in only one centre.

#### 6.6 HANDLING OF MISSING DATA AND OUTLIERS

Data of screened subjects who were withdrawn from the trial prior to first administration of any study drug will not be reported in the CTR.

Data of subjects who failed to complete all periods of the study (dropouts or withdrawals) will be reported in the CTR as far as their data are available. All withdrawals will be documented and the reason for withdrawal recorded in the CTR.

**CTP**: *It is not planned to impute missing values for safety parameters.* 

The only exceptions where imputation might be necessary for safety evaluation are AE dates. Missing or incomplete AE dates are imputed according to BI standards (3).

Missing data and outliers of PK data are handled according to BI standards (4). CTP: PK parameters that cannot be reasonably calculated based on the available drug concentration-time data will not be imputed.

#### 6.7 BASELINE, TIME WINDOWS AND CALCULATED VISITS

Baseline will be defined as the last available value before administration of BI 894416 in period 1 (Visit 2).

Note that this baseline definition will be used for evaluation of data of both treatment periods and of all on-treatment periods ("BI", "ITZ", "BI + ITZ", as defined in <u>Section 6.1</u>).

Time windows are defined in Section 6.1 of the CTP. Adherence to time windows will be checked at the RPM/DBLM.

#### 7. PLANNED ANALYSIS

The format of the listings and tables will follow the BI guideline "Reporting of clinical trials and project summaries" (5).

The individual values of all subjects will be listed. Listings will be sorted by subject number and visit (if visit is applicable in the respective listing). AE listings will be sorted by assigned treatment (see Section 7.8.1 below for details). The listings will be contained in Appendix 16.2 (SDL) of the CTR.

The following standard descriptive statistical parameters will be displayed in summary tables of continuous variables:

N number of non-missing observations

Mean arithmetic mean SD standard deviation

Min minimum Median median Max maximum

For plasma concentrations as well as for all PK parameters the following descriptive statistics will additionally be calculated:

CV arithmetic coefficient of variation

gMean geometric mean

gCV geometric coefficient of variation

For PK parameters the following descriptive statistics will additionally be calculated:

P10 10<sup>th</sup> percentile Q1 1<sup>st</sup> quartile Q3 3<sup>rd</sup> quartile P90 90<sup>th</sup> percentile

The data format for descriptive statistics of plasma concentrations will be identical with the data format of the respective concentrations. The descriptive statistics of PK parameters will be calculated using the individual values with the number of decimal places as provided by the evaluation program. Then the individual values as well as the descriptive statistics will be reported with three significant digits in the CTR.

Tabulations of frequencies for categorical data will include all possible categories and will display the number of observations in a category as well as the percentage (%) relative to the respective treatment group. Percentages will be rounded to one decimal place. The category missing will be displayed if and only if there actually are missing values. Percentages will be based on all subjects in the respective subject set whether they have non-missing values or not.

#### 7.1 DEMOGRAPHIC AND OTHER BASELINE CHARACTERISTICS

Only descriptive statistics are planned for this section of the CTR. These will be based on the TS.

#### 7.2 CONCOMITANT DISEASES AND MEDICATION

Concomitant diseases will be coded according to the most recent version of MedDRA. Concomitant medication will be coded according to the most recent version of the World Health Organisation – Drug Dictionary.

Only descriptive statistics are planned for this section of the CTR.

A medication will be considered concomitant to a treatment, if it

- is ongoing at the time of first administration of the respective treatment or
- starts within the analysis phase of the respective treatment (see <u>Section 6.1</u> for a definition of treatments and analysis phases).

### 7.3 TREATMENT COMPLIANCE

Treatment compliance will not be analysed as a specific endpoint. Any deviations from complete intake will be addressed in the RPM/DBLM (cf. Section 6.2) and described in the CTR.

#### 7.4 PRIMARY ENDPOINT

Analysis of relative bioavailability of primary endpoints  $AUC_{0-tz}$  and  $C_{max}$  of BI 894416 in plasma will be performed as defined in Sections 7.1 and 7.3.1 of the CTP.

The statistical model for the primary analysis defined in the CTP is an analysis of variance (ANOVA) model on the logarithmic scale including "treatment" as fixed effect and "subject" as random effect. In addition, a secondary analysis will be performed, using both, "subject" and "treatment", as fixed effects in the ANOVA model.

Primary PK endpoints will be assessed descriptively. The analysis of standard PK parameters is performed according to BI standards (4) [001-MCS-36-472 RD-01].

#### Exclusion of PK parameters

The ADS ADPP contains column variables APEXC and APEXCO indicating inclusion/exclusion (APEXC) of a PK parameter and an analysis flag comment (APEXCO). All analyses based on the PKS are based on PK parameter values which are not flagged for exclusion, i.e. with APEXC equal to "Included".

#### Exclusion of plasma concentrations

The ADS ADPC (PK concentrations per time-point or per time-interval) contains column variables ACEXC or ACEXCO indicating inclusion/exclusion (ACEXC) of a concentration

and an analysis flag comment (ACEXCO). Exclusion of a concentration depends on the analysis flag comment ACEXCO. For example, if ACEXCO is set to "ALL CALC", the value will be excluded for all types of analyses based on concentrations. If ACEXCO is set to "DESC STATS" the value will be excluded from descriptive evaluations per planned time point/time interval. If ACEXCO contains the addition "TIME VIOLATION" or "TIME DEVIATION", the value can be used for further analyses based on actual times. If ACEXCO is set to "HALF LIFE", the value will be excluded from half-life calculation only; the value is included for all other analyses. Excluded concentration itself will be listed in the CTR associated with an appropriate flag.

Further details are given in "Noncompartmental Pharmacokinetic / Pharmacodynamic Analyses of Clinical Studies" (4) and "Description of Analytical Transfer Files and PK/PD Data Files" (6).

### 7.5 SECONDARY ENDPOINTS

#### 7.5.1 Key secondary endpoint

Not applicable.

#### 7.5.2 Secondary endpoints

Analysis of relative bioavailability of secondary endpoint  $AUC_{0-\infty}$  of BI 894416 in plasma will be performed in the same way as for the primary endpoints.

Additionally, the secondary PK endpoint will be assessed descriptively. The analysis of standard PK parameters is performed according to BI standards (4).

See <u>Section 7.4</u> of this TSAP for details regarding exclusion of PK parameters and plasma concentrations.

#### 7.7 EXTENT OF EXPOSURE

Descriptive statistics are planned for this section of the report.

#### 7.8 SAFETY ANALYSIS

All safety analyses will be performed on the TS.

#### 7.8.1 Adverse events

AEs will be coded with the most recent version of MedDRA.

The analyses of AEs will be descriptive in nature. All analyses of AEs will be based on the number of subjects with AEs and not on the number of AEs.

For analysis, multiple AE occurrence data on the eCRF will be collapsed into one event provided that all of the following applies:

- All AE attributes are identical (lower level term, intensity, action taken, therapy required, seriousness, reason for seriousness, relationship, outcome, AESI)
- The occurrences were time-overlapping or time-adjacent (time-adjacency of two occurrences is given if the second occurrence started at most 1 hour after the first occurrence ended)

For further details on summarization of AE data, please refer to "Analysis and Presentation of Adverse Event Data from Clinical Trials" (7) and "Handling of missing and incomplete AE dates" (3).

The analysis of AEs will be based on the concept of treatment emergent AEs. That means that all AEs will be assigned to the screening or on-treatment phase as defined in <u>Section 6.1</u>. AEs will be analysed based on actual treatments, as defined in <u>Table 6.1: 1</u>.

An overall summary of AEs will be presented. This overall summary will comprise summary statistics for the class of other significant AEs according to ICH E3 (8) and for the class of AESIs.

**CTP:** *The following are considered as AESIs:* 

A hepatic injury is defined by the following alterations of hepatic laboratory parameters:

- o An elevation of AST (aspartate transaminase) and/or ALT (alanine transaminase)  $\geq$ 3-fold ULN combined with an elevation of total bilirubin  $\geq$ 2-fold ULN measured in the same blood sample, or
- Aminotransferase (ALT, and/or AST) elevations  $\geq$ 10 fold ULN

The investigator had to classify on the eCRF whether an observed AE was an AESI or not.

According to ICH E3 (8), AEs classified as "other significant" need to be reported and will include those non-serious and non-significant AEs

(i) which are marked haematological or other lab abnormalities, or

(ii) which were reported with "action taken = discontinuation" or "action taken = reduced", or (iii) which lead to significant concomitant therapy as identified by the Clinical Monitor/Investigator at a Medical Quality Review Meeting.

The frequency of subjects with AEs will be summarised by treatment, primary system organ class (SOC) and preferred term. AEs which were considered by the investigator to be drug related (primary endpoint) will be summarised separately. Separate tables will also be provided for subjects with SAEs, subjects with AESIs and subjects with other significant AEs (according to ICH E3 (8)). The frequency of subjects with AEs and the frequency of subjects with AEs considered by the investigator to be drug related will also be summarised by maximum intensity, primary SOC and preferred term.

The system organ classes and preferred terms within system organ classes will be sorted by descending frequency over all treatment groups.

For disclosure of AE data on ClinicalTrials.gov, the frequency of subjects with non-serious AEs occurring with an incidence of greater than 5 % (in preferred terms) will be summarised by treatment, primary SOC and preferred term. The frequency of subjects with SAEs will also be summarised.

For disclosure of AE data in the EudraCT register, the frequency of AEs, the frequency of non-serious AEs with an incidence of greater than 5 % (in preferred terms) and the frequency of SAEs will be summarised.

For support of lay summaries, the frequency of subjects with drug-related SAEs will be summarised by treatment, primary system organ class and preferred term.

### 7.8.2 Laboratory data

The analyses of laboratory data will be descriptive in nature and will be based on BI standards "Display and Analysis of Laboratory Data" (9).

Analyses will be based on normalised values, which means transforming to a standard unit and a standard reference range. The original values will be analysed if the transformation into standard unit is not possible for a parameter.

Descriptive statistics of laboratory values over time and for the difference from baseline (see Section 6.7) will be provided. Frequency tables of changes between baseline and last value on treatment with respect to the reference range will be presented.

Possibly clinically significant abnormal laboratory values are only those identified either in the Investigator's comments or at the RPM/DBLM at the latest. It is the Investigator's responsibility to decide whether a lab value is clinically significant abnormal or not. Standard or project-specific rules for flagging clinically significant values in an automated manner will not be applied in this study.

Clinically relevant findings in laboratory data will be reported as baseline conditions (at screening) or as AEs (during the trial) if judged clinically relevant by the investigator, and will be analysed as such.

### 7.8.3 Vital signs

The analyses of vital signs (blood pressure and pulse rate) will be descriptive in nature. Descriptive statistics of vital signs over time and for the difference from baseline (see Section 6.7) will be provided.

Clinically relevant findings in vital signs data will be reported as baseline conditions (at screening) or as AEs (during the trial) if judged clinically relevant by the investigator, and will be analysed as such.

#### **7.8.4** Others

Physical and neurological examination findings as well as relevant ECG findings will be reported as relevant medical history/baseline condition (i.e., a condition already existent before intake of first study drug) or as AE and will be summarised as such. No separate listing or analysis of physical or neurological examination as well as ECG findings will be prepared.

TSAP for BI Trial No: 1371-0004 

Proprietary confidential information © 2019 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

#### 8. **REFERENCES**

| 1 | CPMP/ICH/363/96: "Statistical Principles for Clinical Trials", ICH Guideline Topic E9; Note For Guidance on Design, Conduct, Analysis and Evaluation of Clinical Trialss, current version |
|---|---|
| 2 | 001-MCS-40-413_1.0: "Identify and Manage Important Protocol Deviations (iPD)", current version; IDEA for CON |
| 3 | 001-MCG-156_RD-01: "Handling of missing and incomplete AE dates", current version; IDEA for CON |
| 4 | 001-MCS-36-472_RD-01: "Noncompartmental Pharmacokinetic / Pharmacodynamic Analyses of Clinical Studies", current version; IDEA for CON |
| 5 | 001-MCG-159: "Reporting of Clinical Trials and Project Summaries", current version; IDEA for CON |
| 6 | 001-MCS-36-472_RD-03: "Description of Analytical Transfer Files and PK/PD Data Files", current version; IDEA for CON |
| 7 | 001-MCG-156: "Analysis and Presentation of Adverse Event Data from Clinical Trials", current version; IDEA for CON |
| 8 | CPMP/ICH/137/95: "Structure and Content of Clinical Study Reports", ICH Guideline Topic E3; Note For Guidance on Structure and Content of Clinical Study Reports, current version |
| 9 | 001-MCG-157: "Display and Analysis of Laboratory Data", current version; IDEA for CON |

TSAP for BI Trial No: 1371-0004 
Proprietary confidential information © 2019 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

#### **10. HISTORY TABLE**

Table 10: 1 History table

| Version | Date | Author | Sections | Brief description of change |
|---|---|---|---|---|
| | (DD-MMM-YY) | | changed | |
| Final | 06-FEB-2019 | | None | This is the final TSAP without any |
| | | | | modification |